CLINICAL TRIAL: NCT03381196
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Pimodivir in Combination With the Standard-of-care Treatment in Adolescent, Adult, and Elderly Non-hospitalized Subjects With Influenza A Infection Who Are at Risk of Developing Complications
Brief Title: A Study to Evaluate the Efficacy and Safety of Pimodivir in Combination With the Standard-of-Care Treatment in Adolescent, Adult, and Elderly Non-Hospitalized Participants With Influenza A Infection Who Are at Risk of Developing Complications
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on interim Analysis outcome being futile for FLZ3001; decision was taken to stop (early terminate) both FLZ3001/3002. There was no safety concern.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108400; 2017-002217-59 (EudraCT Number); 63623872FLZ3002 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT03834376 (No longer available)
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Influenza A
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (pimodivir + SOC treatment) (Experimental): Participants will receive pimodivir 600 milligram (mg), orally, twice daily, for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of pimodivir on Day 1 [evening], dosing will continue until the morning of Day 6) along with Standard-of-Care (SOC) treatment. The SOC treatment is determined by the investigator based on local practice, and may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of the SOC should be made before randomization. The influenza antiviral should be started no later than Day 2 morning (up to noon). An influenza antiviral as part of the SOC cannot be changed (for example, switching one influenza antiviral for another) during the treatment period, with the exception that an influenza antiviral may be discontinued in the case of a suspected adverse event (AE).
  Interventions: Drug: Pimodivir 600 mg; Other: SOC Treatment
- Treatment Arm 2 (placebo + SOC treatment) (Placebo Comparator): Participants will receive placebo matching to pimodivir orally, twice daily, for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of placebo on Day 1 [evening], dosing will continue until the morning of Day 6) along with SOC treatment. The SOC treatment is determined by the investigator based on local practice, and may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of the SOC should be made before randomization. The influenza antiviral should be started no later than Day 2 morning (up to noon). An influenza antiviral as part of the SOC cannot be changed (for example, switching one influenza antiviral for another) during the treatment period, with the exception that an influenza antiviral may be discontinued in the case of a suspected AE.
  Interventions: Drug: Placebo; Other: SOC Treatment

INTERVENTIONS:
Drug: Pimodivir 600 mg — Participants will receive pimodivir 600 mg, orally, twice daily, for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of pimodivir on Day 1 [evening], dosing will continue until the morning of Day 6).
  Other Names: JNJ-63623872
  Arms: Treatment Arm 1 (pimodivir + SOC treatment)
Drug: Placebo — Participants will receive placebo matching to pimodivir, orally twice daily for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of placebo on Day 1 [evening], dosing will continue until the morning of Day 6).
  Arms: Treatment Arm 2 (placebo + SOC treatment)
Other: SOC Treatment — Participants may receive SOC treatment as a part of background therapy. The SOC treatment is determined by the investigator based on local practice, and may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of the SOC should be made before randomization. The influenza antiviral should be started no later than Day 2 morning (up to noon).

SUMMARY:
The purpose of this study is to evaluate the clinical and virologic benefit of pimodivir in combination with Standard-of-Care (SOC) treatment compared to placebo in combination with SOC treatment.

DETAILED DESCRIPTION:
This double-blind (neither researchers nor participants know what treatment participant is receiving) study will evaluate efficacy/safety of pimodivir in combination with SOC treatment versus placebo in combination with SOC treatment in adolescent (13 to 17 years), adult (18 to 65 years), and elderly (greater than [>] 65 but less than or equal to [<=] 85 years) non-hospitalized participants with influenza A infection who are at risk of developing complications. The study will be conducted in 3 phases: screening phase, double-blind treatment period (5 days), a post treatment follow-up period (23 days). Study evaluations include efficacy, clinical and virological outcomes, pharmacokinetics (PK), PK/pharmacodynamics, biomarkers, safety and tolerability. The duration of participation in the study for each participant is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Present to the clinic with symptoms suggestive of a diagnosis of acute influenza and have at least 1 respiratory symptom and at least 1 systemic symptom, both scored as at least "moderate" if the symptom did not pre-exist before influenza onset, or scored worse than usual if the symptom pre-existed as determined by subject's ratings on Module 1 of the Flu-iiQ and the Pre-existing Symptom Questionnaire in the ePRO device. Symptoms must include the following by category: a) Respiratory symptoms: cough, sore throat, nasal congestion b) Systemic symptoms: headache, body aches or pain, feverishness, fatigue
* Tested positive for influenza A infection after the onset of symptoms, using a rapid influenza diagnostic test (RIDT) or, if available, a polymerase chain reaction (PCR)-based or other rapid molecular diagnostic assay
* Not be in need of hospitalized medical care at screening. Emergency room or hospital observation status for an anticipated duration of less than (<)24 hours is not considered hospitalization as long as a determination of the need for hospitalization has not been made
* Enrollment and initiation of study drug treatment less than or equal to (<=)72 hours after onset of influenza symptoms
* Participants 13 to 65 years of age, inclusive must also have at least 1 of the following: a) Cardiovascular or cerebrovascular disease (including congenital heart disease, chronic heart failure, coronary artery disease, or stroke; excluding isolated hypertension); b) Chronic lung disease (for example, asthma, chronic obstructive lung disease [COPD] or cystic fibrosis); c) Weakened immune system due to disease or medication (for example, participants with human immunodeficiency virus [HIV], cancer, or chronic liver or kidney disease [presence of kidney damage for >3 months, defined by structural or functional abnormalities of the kidney, with or without decreased GFR manifested by: pathological abnormalities; OR markers of kidney damage, including abnormalities in the composition of the blood or urine or abnormalities in imaging tests], or participants taking chronic systemic steroids)

Exclusion Criteria:

* Received more than (>)1 dose of influenza antiviral medication (for example, oseltamivir [OST] or zanamivir), or any dose of ribavirin within 2 weeks, prior to first study drug intake, or received intravenous (IV) peramivir >1 day prior to screening
* Unstable angina pectoris or myocardial infarction within 30 days prior to screening (inclusive)
* Presence of clinically significant heart arrhythmias, uncontrolled, unstable atrial arrhythmia, or sustained ventricular arrhythmia, or risk factors for Torsade de Pointes syndrome
* Known severe hepatic impairment (Child Pugh C cirrhosis) or chronic hepatitis C infection undergoing hepatitis C antiviral therapy
* Severely immunocompromised in the opinion of the investigator (for example, known cluster of differentiation 4 plus [CD4+] count <200 cells per cubic millimeter [cells/mm^3], absolute neutrophil count <750/mm^3, first course of chemotherapy completed within 2 weeks prior to screening, history of stem cell transplant within 1 year prior to screening, history of a lung transplant)

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (427):
- United States (140):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Cahaba Research Inc, Birmingham, Alabama
  - Scottsboro Quick Care Clinic, Scottsboro, Alabama
  - SC Clinical Research Inc., California City, California
  - Research Center of Fresno Inc, Fresno, California
  - Allied Clinical Research, Gold River, California
  - Innovative Clinical Research Inc, Harbor City, California
  - Om Research LLC, Lancaster, California
  - Ark Clinical Research, Long Beach, California
  - Miller Children's Hospital, Long Beach, California
  - Downtown LA Research Center, Inc, Los Angeles, California
  - California Allergy & Asthma Medical Group Inc., Los Angeles, California
  - Adam D. Karns, MD, Los Angeles, California
  - Lucita M. Cruz Md Inc, Norwalk, California
  - Asclepes Research, Panorama City, California
  - Center for Clinical Trials LLC, Paramount, California
  - Benchmark Research, Sacramento, California
  - Medical Associates Research Group, Inc., San Diego, California
  - San Diego Sports Medicine & Family Health Center, San Diego, California
  - West Coast Clinical Research, LLC, San Ramon, California
  - Stanford University, Stanford, California
  - Lynn Institute, Colorado Springs, Colorado
  - Complete Family Care, Northglenn, Colorado
  - Paradigm Clinical Research Centers, Inc., Wheat Ridge, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Moonshine Research Center, Inc, Doral, Florida
  - Best Quality Research Inc, Hialeah, Florida
  - Floridian Clinical Research LLC, Hialeah, Florida
  - The community Research of South Florida, Hialeah, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Homestead Associates in Research Inc, Homestead, Florida
  - Care Partners Clinical Research, Jacksonville, Florida
  - Premier Medical Group, Lady Lake, Florida
  - Sima Research Clinic, Miami, Florida
  - Universal Clinical Research Associates, Miami, Florida
  - South Florida Research Center Inc., Miami, Florida
  - A Plus Research, Miami, Florida
  - Nuren Medical & Research Center, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Combined Research Orlando, Orlando, Florida
  - Clinical NeuroScience Solutions Inc, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - Pines Care Research Center Inc, Pembroke Pines, Florida
  - South Broward Research, LLC, Pembroke Pines, Florida
  - Destin Pulmonary Critical Care, PLLS., Santa Rosa Beach, Florida
  - Vita Health and Medical center, Tamarac, Florida
  - Asclepes Research, Weeki Wachee, Florida
  - Axcess Medical Research, LLC, Wellington, Florida
  - Cozy Research, Llc, Zephyrhills, Florida
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Saltzer Medical Group, Nampa, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Medisphere Medical Research Center, Llc, Evansville, Indiana
  - Hutchinson Clinic, Hutchinson, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Medpharmics, LLC, Metairie, Louisiana
  - North Star Clinical Research, LLC, Shreveport, Louisiana
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State Univ School of Medicine, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Tri County Research, Inc., Sterling Heights, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Arcturus Healthcare PLC, Troy, Michigan
  - Craig A. Spiegel, MD, Bridgeton, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Montana Medical Research, Missoula, Montana
  - Barrett Clinic P.C., La Vista, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Next Phase Research Alliance, Las Vegas, Nevada
  - Saint Michaels Medical Center, Newark, New Jersey
  - Accellacare Research of Cary, Cary, North Carolina
  - Onsite Clinical Solutions, Clemmons, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - clinical research of Gastonia, Gastonia, North Carolina
  - Hickory Research Center., Hickory, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Clinical Trials of America, Winston-Salem, North Carolina
  - Southeastern Research Center LLC, Winston-Salem, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Buckeye Health and Research, LLC, Hilliard, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Detweiler Family Medicine and Associates, Lansdale, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians Research, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians Research, Uniontown, Pennsylvania
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - Spectrum Medical Research, Gaffney, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Fusion Clinical Research of Spartanburg, Spartanburg, South Carolina
  - Invocare Clinical Research Center, West Columbia, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - PMG Research of Bristol, Bristol, Tennessee
  - PMG Research of Knoxville, Jefferson City, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - HIRG, LLC dba Health Innovation Research Group, Arlington, Texas
  - ACRC Trials, Austin, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - WR-Global Medical Research, LLC, DeSoto, Texas
  - University Of Texas Medical Branch At Galveston, Galveston, Texas
  - San Gabriel Clinical Research, LLC, Georgetown, Texas
  - BI Research Center, Houston, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - Northwest Med Care,P.A., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Dairy Ashford Family Practice, Houston, Texas
  - JM Research.PLLC, Houston, Texas
  - PCP for Life, Houston, Texas
  - SMS Clinical Research LLC, Mesquite, Texas
  - Village Health Partners, Plano, Texas
  - Tekton Research Inc., San Antonio, Texas
  - DM Clinical Research, San Antonio, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Val Hansen, Bountiful, Utah
  - Ericksen Research and Development, Clinton, Utah
  - J. Lewis research Inc./ Foothill Family Clinic South, Draper, Utah
  - Advanced Research Institute, Ogden, Utah
  - Granger Medical Clinic-Riverton, Riverton, Utah
  - J. Lewis research Inc./ Foothill Family Care, Salt Lake City, Utah
  - J. Lewis research Inc./ Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research Inc/ FirstMed East, Salt Lake City, Utah
  - J. Lewis Research Inc./Jordan River Family Medicine, South Jordan, Utah
  - Millennium Clinical Trials LLC, Arlington, Virginia
- Argentina (14):
  - Hospital Interzonal General de Agudos Dr. Jose Penna, Bahía Blanca
  - CEMIC Saavedra, Ciudad de Buenos Aires
  - Hospital Nuestra Señora de la Misericordia, Córdoba
  - Hospital Rawson, Córdoba
  - Hospital San Roque, Córdoba
  - Sanatorio Allende, Córdoba
  - Hospital Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Sanatorio Juan XXIII, General Roca
  - Sanatorio del Oeste Ituzaingo, Ituzaingó
  - Instituto Medico Platense, La Plata
  - Hospital Italiano de La Plata, La Plata Lpl Lpl
  - Sanatorio Britanico S.A., Rosario
  - Instituto Del Buen Aire, Santa Fe
- Australia (2):
  - Northside Health, Coffs Harbour
  - Mater Hospital Brisbane, South Brisbane
- Austria (2):
  - AKH - Medizinische Universitat Wien, Vienna
  - SMZ Süd - Kaiser Franz Josef Spital Wien, Vienna
- Belgium (9):
  - CHU Saint-Pierre, Brussels
  - Hopital Erasme, Brussels
  - Institut Jules Bordet, Brussels
  - De Meulemeester, Marc, Gozée
  - Jaak Mortelmans, Ham
  - Quartier du Furgy 4, Herbeumont
  - Research Link, Linkebeek
  - BVBA Dr. Luc Capiau, Massemen
  - Testumed, Tessenderlo
- Brazil (13):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Infection Control Ltda, Brasil
  - Hrpc Ulbratech - Ulbra, Canoas
  - Centro de Estudos Clínicos do Interior Paulista - CECIP, Jaú
  - CMIP - Centro Mineiro de Pesquisa Ltda, Juiz de Fora
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - CCBR Brasil Centro de Pesquisas e Análises Clínicas Ltda., Rio de Janeiro
  - Pesquisare Saude, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Fundacao Jose Luiz Egydio Setubal, São Paulo
- Bulgaria (10):
  - SHATPPD - Ruse Ltd., Rousse
  - MHAT Knyaginya Klementina, Sofia
  - MHAT 'Lyulin' EAD, Sofia
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - DCC II- Sofia EOOD, Sofia
  - Medical Center 'N. I. Pirogov', EOOD, Sofia
  - Medical Center Excelsior OOD, Sofia
  - Military Medical Academy - Sofia, Sofia
  - MHAT Dr Stefan Cherkezov, Veliko Tarnovo
  - MC 'Sv. Ivan Rilski', OOD, Vidin
- Canada (7):
  - The Bailey Clinic, Red Deer, Alberta
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Aggarwal and associates Ltd, Brampton, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Dr. Anil K Gupta Medicine Professional Corporation, Toronto, Ontario
  - Recherche Clinique Sigma Inc., Québec, Quebec
- Chile (3):
  - Hospital El Pino, San Bernardo
  - Centro de Investigacion del Maule, Talca
  - Hospital de Niños y Cunas, Viña
- China (5):
  - Chinese PLA General Hospital, Beijing
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Wuxi People s Hospital, Wuxi
  - Henan Provincial Peoples Hospital, Zhengzhou
- Czechia (6):
  - ADMED s.r.o., České Budějovice
  - Sanare, s.r.o., České Budějovice
  - Nemocnice Kyjov, p.o., Kyjov
  - Praktik Pb s.r.o, Příbram
  - SARKAMED s.r.o., Slaný
  - Prakticky lekar, Sokolov
- Estonia (6):
  - Private GP Ilme Last, Paide
  - Vee Family Doctor's Center OY, Paide
  - OU Innomedica, Tallinn
  - Merelahe Family Doctors Center, Tallinn
  - Pirita Family Doctors Centre, Tallinn
  - Family Doctors Pullerits & Gavronski, Tartu
- France (8):
  - Centre Hospitalier d'Agen, Agen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Départemental, La Roche S/ Yon Cedex 9
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - CHU Nantes - Hotel Dieu, Nantes
  - CHU De Nice Hopital De l'Archet, Nice
  - Hôpital Bichat - Claude Bernard, Paris
  - Hopital Cochin, Paris
- Germany (7):
  - Universitaetsklinikum Koelnt, Cologne
  - MECS GmbH Cottbus, Cottbus
  - Jung, Thomas, Deggingen
  - Universitaetsklinik Erlangen, Erlangen
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Gemeinschaftspraxis Dr. Klein/ Minnich, Künzing
  - Gemeinschaftspraxis Dr. Taeschner / Dr. Bonigut, Leipzig
- Hungary (15):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Eszak Kozep budai Centrum Uj Szent Janos Korhaz es Szakrendelo Budai Csaladkozpontu, Budapest
  - Strázsahegy Medicina Bt, Budapest
  - Pestszentimrei Gyermekrendelő, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Futurenest Klinikai Kutato Kft., Miskolc
  - Mohacsi Korhaz, Mohács
  - Borbanya Praxis Eu. Kft., Nyíregyháza
  - Medifarma-98 Kft., Nyíregyháza
  - DRC Szentendre, Szentendre
  - Tudogyogyintezet Torokbalint, Törökbálint
  - DRC Zamardi, Zamárdi
  - DRC Zirc, Zirc
- India (14):
  - Rajiv Gandhi Institute of Medical Sciences, Balaga
  - M S Ramaiah Memorial Hospital, Bangalore
  - S. R. Kalla Memorial General Hospital, Jaipur
  - Midland Healthcare & Research Center, Lucknow
  - Kasturba Medical College Hospital, Manipal
  - Suretech Hospital and Research Centre Limited, Nagpur
  - Siddhi Hospital, Nashik
  - BLK Super Specialty Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Sahyadri Speciality Hospital, Pune
  - Lifepoint Multispecialty Hospital, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Unique Hospital, Surat
  - BAPS Pramukhswami Hospital, Surat
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
- Italy (4):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Policlinico di Modena, Modena
  - Azienda Socio Sanitaria Territoriale di Monza Presidio San Gerardo, Monza
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Latvia (11):
  - Liga Kozlovska family doctor practice, Balvi
  - OLVI Medical Centre, Daugavpils
  - Baiba Bake GP practice, Jelgava
  - Ruta Eglite's Private Practice, Kuldīga
  - Inese Cebere GP practice, Liepāja
  - S. Boreiko Doctor's Practice, Ogre
  - Children's Clinical University Hospital, Riga
  - Clinic of GP A.Lasmanis 'ALMA', Riga
  - Health Centre 4, Riga
  - Inese Petrova General Practitioner Practice, Tukums
  - Medical Practice BINI, Ventspils
- Lithuania (9):
  - Auki Sveikas, Kaunas
  - Silainiai Family Health Center, JSC, Kaunas
  - Saules Seimos Medicinos Centras, JSC, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Inlita, JSC, Lazdynai KTC clinical trial site, Vilnius
  - Central Outpatient Clinic, Vilnius
  - Inlita, JSC, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Public Institution, Vilnius
- Malaysia (4):
  - Klinik Kesihatan Cheras Baru, Cheras Baru
  - Klinik Kesihatan Kuang, Kuang
  - Hospital Miri, Miri
  - Hospital Taiping, Taiping
- Mexico (9):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada S.C., Culiacán
  - Centro de Investigacion Medico Biologica y Terapia Avanzada CIMBYTA, Guadalajara
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara
  - Centro Medico Jojutla, Jojutla
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Hospital Universitario de Nuevo Leon 'Dr Jose Eleuterio Gonzalez', Monterrey
  - Clinical Trials Mexico S.A. de C.V., Pahucha
- Netherlands (3):
  - Huisartsenpraktijk Zijtregtop, Rotterdam
  - Huisartsenpraktijk Mangal, The Hague
  - Huisartsenpraktijk Top, Zwijndrecht
- New Zealand (4):
  - Southern Clinical Trials Ltd, Auckland
  - Culloden Research Ltd, Papamoa
  - Lakeland Family Medical Services Ltd, Rotorua
  - Wellington Hospital, Wellington
- Peru (5):
  - Complejo Hospitalario San Pablo, Lima
  - Clínica Sanna San Borja, Lima
  - Clínica Internacional, Lima
  - Hospital Maria Auxiliadora, Lima
  - Clinica Peruano Americana S.A, Trujillo
- Poland (6):
  - Malopolskie Centrum Alergologii, Krakow
  - ETG Lodz, Lodz
  - Powiatowe Centrum Medyczne w Wolowie Sp z o o, Specjalistyczna W Brzegu Dolnym
  - Gabinet Lekarski Pediatryczno-Alergologiczny, Sucha Beskidzka
  - NZOZ Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Centrum Medyczne w Lancucie Sp.z o.o., Łańcut
- Russia (10):
  - Institute Of Epidimiology And Microbiology, Kazan'
  - Limited Liability company 'MSMC' Euromed, Omsk
  - LLC Outpatient department of Private Security Guards and Detectives, Saint Petersburg
  - LLC Institute of Medical Examinations, Saint Petersburg
  - LLC Kurator, Saint Petersburg
  - FSBI 'Scientific and Research Institute of Flu' of the MoH of the RF, Saint Petersburg
  - LLC 'ArsVite', Stavropol
  - Siberian State Medical University, Tomsk
  - Clinical Hospital #3, Yaroslavl
  - SBEI HPE 'Yaroslavl State Medical University' of the MoH of the RF, Yaroslavl
- Slovakia (4):
  - Alersa, S.R.O., Košice
  - Nemocnica s poliklinikou S. Kukuru Michalovce, a.s., Michalovce
  - Plucna ambulancia Hrebenar, s.r.o., Spišská Nová Ves
  - Nemocnica arm. generala L. Svobodu Svidnik, a.s.,, Svidník
- South Africa (34):
  - Cardiology Clinical Research, Alberton
  - Josha Research, Bloemfontein
  - Dr Dindar & Partner, Breyten
  - Endocare Research, Cape Town
  - Uhuru Clinical Trial Centre, Cape Town
  - Dr EL Janari Private Practice, Cape Town
  - Precise Clinical Solutions, Chatsworth
  - Abdullah, IA, Durban
  - Sebastian, Peter, Durban
  - Pillai, P, Durban
  - Govind, U, Durban
  - Jeevren Reddy, MD, Durban
  - Global Clinical Research SA, Durban North
  - CRISMO Bertha Gxowa Research Centre, Johannesburg
  - Peermed Clinical Trial Centre, Kempton Park
  - DJW Research, Krugersdorp
  - Aliwal Shoal Medical Centre, KwaZulu-Natal
  - Dr A Jacovides Clinical Trials Inc., Midrand
  - Dr AA Mahomed Medical Centre, Moloto South
  - Newtown Clinical Research, Newtown
  - Pillay, SR, Ottawa
  - Smartmed Research Centre, Port Elizabeth
  - Emmed Research, Pretoria
  - Botho ke Bontle Health Services, Pretoria
  - Into Research, Pretoria
  - Jongaie Research, Pretoria
  - Queenswood Clinical Trial Centre, Pretoria
  - Engelbrecht, I, Pretoria
  - Johese Clinical Research, Pretoria
  - Wits Clinical Research, Soweto
  - Limpopo Clinical Research Initiative, Thabazimbi
  - Clinteam Vaal Clinical Trial Centre, Van Der Bijl
  - Welkom Clinical Trial Centre, Welkom
  - Moriana Clinical Research, Winnie Mandela
- South Korea (13):
  - Chungbuk National University Hospital, Cheongju-si
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Inha University Hospital, Incheon
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Dong-A University Hospital, Pusan
  - Korea University Anam Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic university of Korea ST Vincent Hospital, Suwon
- Spain (10):
  - Hosp. Gral. Univ. de Elche, Elche
  - Hosp. Univ. San Cecilio, Granada
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (4):
  - Department for Heart Failure and Valvular Disease, Malmo
  - City Diabetes, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (5):
  - Taipei Medical University Shuang-Ho Hospital, New Taipei City
  - Kuang Tien General Hospital, Shalu, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Medical University-Wan Fang Hospital, Taipei
- Thailand (5):
  - The Hospital for Tropical Diseases, Bangkok
  - Siriraj Hospital, Bangkok
  - Srinagarind Hospital, Muang
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi
  - Bumrungrad Hospital, Wattana
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty, Ankara
  - Adnan Menderes University, Aydin
  - Uludag University Medical Faculty, Bursa
  - Diyarbakir University Medical Faculty, Diyarbakır
  - Kocaeli University Medical Faculty, Kocaeli
  - Hacettepe University Medical Faculty, Samanpazarı
  - Karadeniz Teknik University Medical Faculty, Trabzon
- Ukraine (5):
  - Med San Unit OJSC Kharkiv S.OrdzhonikidzeTractor Plant Dept of Ther KMA PGE, Kharkiv
  - Kyiv Oleksandrivska Clinical Hospital, Kyiv
  - Odesa City Municipal Institution Polyclinic #20, Odesa
  - Poltava Regional Clinical Hospital HSEI of Ukraine Ukrainian Medical Stomatological Academy, Poltava
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
- United Kingdom (5):
  - Swan Lane Medical Centre, Bolton
  - Bodey Medical Centre, Manchester
  - Barlow Medical Centre, Manchester
  - West Timperley Medical Centre, Manchester
  - Northenden Group Practice, Northenden
- Vietnam (3):
  - Bach Mai Hospital, Hanoi
  - National Hospital for Tropical Diseases, Hanoi
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Leopold L, Vingerhoets J, Deleu S, Nalpas C, Weber K, van Dromme I, Lowson D, Michiels B, van Duijnhoven W. Efficacy and Safety of Pimodivir Combined With Standard of Care in Hospitalized and Nonhospitalized High-Risk Adolescents and Adults With Influenza A Infection. J Infect Dis. 2025 Feb 4;231(1):e132-e143. doi: 10.1093/infdis/jiae408. PMID 39172627

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimodivir + SOC: Participants received 600 milligrams (mg) pimodivir twice daily (bid) on Day 1 through Day 5 along with standard of care (SOC) treatment.
- Placebo + SOC: Participants received matching placebo bid on Day 1 through Day 5 along with SOC treatment.
Period: Overall Study
Arm/Group | Pimodivir + SOC | Placebo + SOC
Started | 276 | 277
Treated | 273 | 271
Completed | 260 | 258
Not Completed | 16 | 19
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Other | 0 | 1
Not completed — Lost to Follow-up | 5 | 4
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Randomized, not treated | 3 | 6

BASELINE CHARACTERISTICS:
Population: The safety set (or all participants treated) includes all participants who received at least one dose of study drug and were analyzed by treatment arm as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimodivir + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 273 | 271 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (16.6) | 50.3 (17.35) | 50.7 (16.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 141 | 293
  Male | 121 | 130 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 89 | 172
  Not Hispanic or Latino | 185 | 178 | 363
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 27 | 34 | 61
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 33 | 28 | 61
  White | 206 | 201 | 407
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 13 | 12 | 25
  AUSTRALIA | 2 | 1 | 3
  BELGIUM | 3 | 1 | 4
  BRAZIL | 1 | 0 | 1
  BULGARIA | 8 | 2 | 10
  CANADA | 1 | 3 | 4
  ESTONIA | 0 | 1 | 1
  FRANCE | 1 | 1 | 2
  GERMANY | 2 | 2 | 4
  HUNGARY | 1 | 1 | 2
  INDIA | 5 | 3 | 8
  ITALY | 0 | 3 | 3
  LATVIA | 1 | 0 | 1
  LITHUANIA | 6 | 5 | 11
  MALAYSIA | 1 | 0 | 1
  MEXICO | 3 | 4 | 7
  POLAND | 1 | 2 | 3
  RUSSIAN FEDERATION | 1 | 1 | 2
  SOUTH AFRICA | 25 | 33 | 58
  SOUTH KOREA | 0 | 2 | 2
  SPAIN | 1 | 1 | 2
  SWEDEN | 1 | 0 | 1
  TAIWAN | 2 | 4 | 6
  THAILAND | 8 | 5 | 13
  TURKEY | 2 | 2 | 4
  UKRAINE | 6 | 4 | 10
  UNITED KINGDOM | 0 | 1 | 1
  UNITED STATES | 178 | 177 | 355

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of 7 Primary Influenza-related Symptoms as Assessed by the Patient-Reported Outcome (PRO) Measure Flu-Intensity and Impact Questionnaire (Flu-iiQ)
Description: The Flu-iiQ is a PRO that measures influenza symptom intensity (none, mild, moderate, or severe) on a 4 point Likert response rating scale ranging from 0 to 3, where "0" represents the absence of symptom and "3" represents the severe symptom. The resolution of influenza-related symptoms is defined as the beginning of the 24-hour period that 7 influenza symptoms (cough, sore throat, headache, nasal congestion, feeling feverish, body aches and pains, fatigue) are at most mild or at least back to previous level of symptom severity in case the participant reported the symptom as pre-existing.
Time Frame: Up to Day 28
Population: The Intent-To-Treat infected (ITT-i) Set included all randomized participants who received at least 1 dose of study drug and who had confirmed infection with influenza A and analyzed by planned treatment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 223 | 223
hours | 92.62 [77.60 to 104.20] | 105.13 [92.73 to 128.63]
Statistical Analysis 1: Comparison: Pimodivir + SOC vs Placebo + SOC; Test type: Superiority; p = 0.0216, Gehan-Wilcoxon test

2. Secondary Outcome: Number of Participants Hospitalized After Treatment Initiation
Description: The number of participants hospitalized after treatment initiation were reported.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 223 | 223
Participants | 4 | 4

3. Secondary Outcome: Viral Load Over Time
Description: Viral load over time was measured by quantitative real time polymerase chain reaction (qRT-PCR) and viral culture in the mid-turbinate (MT) nasal swabs and endotracheal samples.
Time Frame: Baseline, Day 3, 6, 10, 14
Population: The Intent-To-Treat infected (ITT-i) Set included all randomized participants who received at least 1 dose of study drug and who had confirmed infection with influenza A and analyzed by planned treatment. Here N (number of participants analyzed) are participants evaluable for this outcome measure and "n (number analyzed)" signifies number of participants analyzed for specified categories.
Measure: Mean (Standard Deviation); unit: log 10 viral particles per milliliter
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 221 | 216
log 10 viral particles per milliliter
  Baseline | 5.891 (1.5745) | 5.914 (1.4947)
  Day 3: number analyzed (Participants) | 203 | 210
  Day 3 | 3.558 (1.1918) | 4.244 (1.3535)
  Day 6: number analyzed (Participants) | 206 | 210
  Day 6 | 2.644 (0.9159) | 2.833 (1.0432)
  Day 10: number analyzed (Participants) | 203 | 211
  Day 10 | 2.234 (0.4586) | 2.289 (0.6279)
  Day 14: number analyzed (Participants) | 206 | 209
  Day 14 | 2.153 (0.3904) | 2.162 (0.4355)

4. Secondary Outcome: Number of Participants With Emergence of Viral Resistance to Pimodivir
Description: Emergence of viral resistance to pimodivir was detected by genotyping and/or phenotyping. Nasal MT swabs and endotracheal samples were used for sequence analysis of the polymerase basic protein (PB)2 region of the influenza polymerase gene, and of neuraminidase (NA) genes for participants using an NA inhibitor (NAI) as part of their Standard of Care (SOC).
Time Frame: Up to Day 28
Population: Population included participants from ITT-i set with both baseline and post-baseline sequencing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 71 | 108
Participants | 4 | 0

5. Secondary Outcome: Plasma Concentration of Pimodivir
Description: Plasma concentration of Pimodivir was reported.
Time Frame: Day 3, 6, 7
Population: The Safety Set (or all participants treated) included all participants who received at least one dose of study drug and were analyzed by treatment arm as treated. Here, N (number of participants analyzed) signifies participants evaluable for this outcome measure and "n (number analyzed)" signifies number of participants analyzed for specified categories.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Pimodivir + SOC
Number analyzed (Participants) | 200
nanograms per milliliter (ng/mL)
  Day 3 | 1233.0 (1912.6)
  Day 6: number analyzed (Participants) | 180
  Day 6 | 933.8 (2131.4)
  Day 7: number analyzed (Participants) | 45
  Day 7 | 276.7 (308.6)

6. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to Day 28
Population: The Safety Set (or all participants treated) included all participants who received at least one dose of study drug and were analyzed by treatment arm as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 273 | 271
Participants | 123 | 101

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Tests
Description: Number of participants with clinically significant changes in laboratory tests were reported. Blood samples for hematology, serum chemistry, and urinalysis was collected at predefined time points for clinical laboratory testing.
Time Frame: Up to Day 28
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 273 | 271
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG)
Description: Number of participants with clinically significant changes in Electrocardiogram (ECG) were reported.
Time Frame: Up to Day 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 273 | 271
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants with clinically significant changes in vital signs (temperature, pulse rate, respiratory rate and blood pressure) were reported.
Time Frame: Up to Day 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 273 | 271
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: The Safety Set (or all participants treated) included all participants who received at least one dose of study drug and were analyzed by treatment arm as treated.
Arm/Group | Pimodivir + SOC | Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 0/273 | 1/271
Serious Adverse Events (participants affected / at risk) | 3/273 | 4/271
Other Adverse Events (participants affected / at risk) | 122/273 | 99/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimodivir + SOC (N=273) | Placebo + SOC (N=271)
Bacteraemia (Infections and infestations) | 0 | 1
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Streptococcal Sepsis (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimodivir + SOC (N=273) | Placebo + SOC (N=271)
Neutropenia (Blood and lymphatic system disorders) | 3 | 7
Polycythaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 1
Conjunctival Haemorrhage (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 54 | 18
Faeces Soft (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Infrequent Bowel Movements (Gastrointestinal disorders) | 0 | 1
Lip Disorder (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 10
Pancreatic Atrophy (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 9
Fatigue (General disorders) | 3 | 0
Feeling Jittery (General disorders) | 0 | 1
Impaired Healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Peripheral Swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 4
Vessel Puncture Site Bruise (General disorders) | 0 | 2
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 2
Abscess (Infections and infestations) | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1
Adenoviral Upper Respiratory Infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 7 | 9
Bronchitis Bacterial (Infections and infestations) | 0 | 2
Candida Infection (Infections and infestations) | 0 | 1
Ear Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Kidney Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0
Oral Candidiasis (Infections and infestations) | 1 | 1
Otitis Externa (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Otitis Media Acute (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 7 | 4
Skin Candida (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 11 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 4
Amylase Abnormal (Investigations) | 1 | 0
Amylase Increased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 1
Blood Bilirubin (Investigations) | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 3 | 3
Blood Glucose Increased (Investigations) | 1 | 0
Blood Potassium Increased (Investigations) | 3 | 0
Blood Pressure Decreased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 1
Glomerular Filtration Rate Decreased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 1
International Normalised Ratio Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 1
Pancreatic Enzymes Increased (Investigations) | 2 | 1
Transaminases Increased (Investigations) | 2 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 2 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Intercostal Neuralgia (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal Pain (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 2
Hot Flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
As the study was terminated early after a pre-planned interim analysis which showed futility, the Sponsor decided not to perform the complete analysis planned per protocol. Hence, data was collected and analyzed for safety and selected efficacy parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03381196/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03381196/SAP_001.pdf